CLINICAL TRIAL: NCT03948620
Title: Associations Between Macrolide Antibiotics Prescribed During Pregnancy and Adverse Child Outcomes
Brief Title: Macrolide in Pregnancy and Adverse Child Outcomes
Status: Completed | Type: Observational
Sponsor: Institute of Child Health (Other)
Responsible Party: Sponsor
Other Study IDs: Heng1
Record Dates: First submitted 2019-05-10; First posted 2019-05-14 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Infection
MeSH Terms: conditions — Infections | interventions — Macrolides; Penicillins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children whose mother prescribed antibiotics during pregnancy: Children whose mother were prescribed an only monotherapy of macrolides or penicillins from 5 gestational weeks (GW) to delivery. A monotherapy is defined as one or more consecutive prescriptions for a single antibiotic (i.e. same drug substance) separated by no more than 30 days and uninterrupted by prescriptions for other antibiotic drug substances.
  The investigators will also build a negative control cohort which includes children whose mother were prescribed an only monotherapy of macrolides or penicillins from 50 to 10 weeks before conception.
  Interventions: Drug: Macrolides; Drug: Penicillins

INTERVENTIONS:
Drug: Macrolides — Macrolide antibiotics, including erythromycin, clarithromycin and azithromycin. Prescriptions of macrolides will be identified using a drug code list based on the British National Formulary (chapter 5.1.5) and the date of the first prescription was used as the index date of exposure.
Drug: Penicillins — The comparison group consists of children whose mother were prescribed penicillins during pregnancy. Prescriptions of penicillins will be identified using a drug code list based on the British National Formulary (chapter 5.1.1) and the date of the first prescription will be used as the index date of exposure.

SUMMARY:
Over the last 20 years, concerns have been raised about rare but serious adverse outcomes associated with macrolide use during pregnancy. The strongest evidence comes from a large randomised controlled trial (RCT, ORACLE Child Study II) of women with spontaneous preterm labour (SPL), which reported an increased risk of cerebral palsy in children whose mothers received erythromycin compared with no erythromycin. A recent systematic review on macrolides prescription during pregnancy showed consistent associations with miscarriage, and less consistent associations with adverse child outcomes such as congenital malformations, cerebral palsy and epilepsy. In this study, the investigators will evaluate associations between macrolide antibiotics prescription during pregnancy and a range of adverse child outcomes.

The investigators compare children whose mothers were prescribed an only monotherapy of macrolides or penicillins during pregnancy (from 5 gestational week (GW) to delivery and by trimesters). The investigators estimate the risk ratios of major malformation (overall and five system-specific) and hazard ratios of four neurodevelopmental disorders (cerebral palsy, epilepsy, attention-deficit/hyperactivity disorder, and autism spectrum disorder) with control for potential confounders. The associations will also be examined by subtype of macrolides and treatment duration.

Mother-child pairs will be analysed in a cohort selected from the UK Clinical Practice Research Database (CPRD) between 1990 and 2016.

ELIGIBILITY:
Inclusion Criteria:

* Children whose mother was prescribed an only monotherapy of macrolides or penicillins during pregnancy (between 5 GW and delivery).
* Children born from Jan 1st 1990 to June 30th 2016 in the CPRD Mother Baby Link.
* Children who registered with the GP within 6 months of birth
* Children whose mother was aged 14 to 50 years and had been registered with GP at least 50 weeks before estimated conception date until after delivery

Exclusion Criteria:

* Children with known chromosomal abnormalities and pregnancies with exposure to known teratogenic medications (warfarin, angiotensin-converting enzyme (ACE) inhibitors, antineoplastic agents, isotretinoin, misoprostol, and thalidomide)

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will consist of all eligible children from the source population where the mother was prescribed an only monotherapy of macrolides or penicillins during pregnancy. The source population will be all mother-baby pairs identified from CPRD Mother-baby linkage where the children were born from Jan 1st 1990 to June 30th 2016.
Sampling Method: Probability Sample
Enrollment: 726274 (Actual)
Dates: Start 1990-01-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Number of major malformation overall | From birth up to 4 years after birth.
  Major malformation overall will be defined as any of the 11 major system-specific malformations defined in the European Surveillance of Congenital Anomalies (EUROCAT)(Congenital heart defect, nervous system, eye, ear/face/neck, respiratory tract, oro-facial cleft, digestive system, abdominal wall defect, urinary tract, genital tract, and other malformations). The investigators exclude musculoskeletal malformations which are not reliably recorded in general practice (GP) records, and malformation with known cause such as malformation resulted from maternal infections, fetal alcohol syndrome and chromosomal malformations. The malformations will be identified in the children's medical records using Read codes mapped from the tenth edition of the International Classification of Diseases (ICD-10) code lists provided by EUROCAT.
Number of cardiovascular malformation | From birth up to 4 years after birth.
  The malformations will be identified in the children's medical records using Read codes mapped from the tenth edition of the International Classification of Diseases (ICD-10) code lists provided by EUROCAT (ICD Q20-Q26; exclude Q2111, Q250 if gestational age (GA) <37 weeks, Q2541, Q256 if GA<37 weeks, and Q261).
Number of nervous system malformation | From birth up to 4 years after birth.
  The malformations will be identified in the children's medical records using Read codes mapped from the tenth edition of the International Classification of Diseases (ICD-10) code lists provided by EUROCAT (Q00-Q07, exclude Q0461, Q0782).
Number of gastrointestinal system malformation | From birth up to 4 years after birth.
  The malformations will be identified in the children's medical records using Read codes mapped from the tenth edition of the International Classification of Diseases (ICD-10) code lists provided by EUROCAT (Q38-Q45, Q790, exclude Q381, Q382, Q3850, Q400, Q401, Q4021, Q430, Q4320, Q4381, Q4382).
Number of genital malformation | From birth up to 4 years after birth.
  The malformations will be identified in the children's medical records using Read codes mapped from the tenth edition of the International Classification of Diseases (ICD-10) code lists provided by EUROCAT (Q50-Q52, Q54-Q56; exclude Q523, Q525, Q527, Q5520, Q5521).
Number of urinary malformation | From birth up to 4 years after birth.
  The malformations will be identified in the children's medical records using Read codes mapped from the tenth edition of the International Classification of Diseases (ICD-10) code lists provided by EUROCAT (Q60-Q64, Q794; exclude Q610, Q627, Q633).
Rate of cerebral palsy | From birth up to 15 years after birth.
  The investigators identify children with cerebral palsy using informative Read codes or prescription codes (selected by the Random Forest approach) and validated by a paediatric neurologist (FC) and a clinical epidemiologist with paediatrics expertise (RG) blinded to their prenatal exposure (A machine learning approach to identify cases of cerebral palsy using the UK primary care database.Fan, Heng et al.The Lancet , Volume 392 , S33).
Rate of epilepsy | From birth up to 15 years after birth.
  The investigators identify epilepsy by 2 prescriptions of antiepileptic drug (AED, identified based on British National Formula Chapter 4.8) within 4 months or >= 1 diagnosis in children's GP records.
Rate of attention-deficit/hyperactivity disorder (ADHD) | From birth up to 15 years after birth.
  The investigators identify ADHD by >= 2 occurrence of prescriptions for ADHD ( identified based on British National Formula Chapter 4.4) or diagnoses (attention deficit hyperactivity disorder, hyperkinetic disorders, hyperkinetic syndrome, hyperkinetic reaction of childhood or adolescence, overactive child syndrome and disturbance of activity and attention) in children's GP records.
Rate of autism spectrum disorder (ASD) | From birth up to 15 years after birth.
  The investigators identify ASD by at least 1 diagnostic code ((infantile or childhood) autism, Asperger's syndrome, Rett's syndrome, Heller's syndrome, Autistic spectrum disorder, disintegrative disorder, and other pervasive developmental disorders) in children's GP records.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Gilbert, MD, Study Director — Institute of Child Health, University College London; Leah Li, PhD, Study Director — Institute of Child Health, University College London

REFERENCES:
- [Background] Kenyon S, Pike K, Jones DR, Brocklehurst P, Marlow N, Salt A, Taylor DJ. Childhood outcomes after prescription of antibiotics to pregnant women with spontaneous preterm labour: 7-year follow-up of the ORACLE II trial. Lancet. 2008 Oct 11;372(9646):1319-27. doi: 10.1016/S0140-6736(08)61203-9. Epub 2008 Sep 17. PMID 18804276
- [Background] Fan H, Li L, Wijlaars L, Gilbert RE. Associations between use of macrolide antibiotics during pregnancy and adverse child outcomes: A systematic review and meta-analysis. PLoS One. 2019 Feb 19;14(2):e0212212. doi: 10.1371/journal.pone.0212212. eCollection 2019. PMID 30779772
- [Derived] Fan H, Gilbert R, O'Callaghan F, Li L. Associations between macrolide antibiotics prescribing during pregnancy and adverse child outcomes in the UK: population based cohort study. BMJ. 2020 Feb 19;368:m331. doi: 10.1136/bmj.m331. PMID 32075790

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-22): https://cdn.clinicaltrials.gov/large-docs/20/NCT03948620/Prot_SAP_000.pdf